CLINICAL TRIAL: NCT04813276
Title: Efficacy of a Self-advocacy Serious Game Intervention for Women With Advanced Cancer
Brief Title: Efficacy of a Self-advocacy Serious Game Intervention
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Teresa Thomas, PhD, RN, Assistant Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: STUDY21020095
Record Dates: First submitted 2021-03-20; First posted 2021-03-24 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Self-Management; Quality of Life
Keywords: Self-advocacy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Serious game intervention (Experimental): Participants receive the Strong Together serious game program on a tablet computer.
  Interventions: Behavioral: Strong Together serious game
- Enhanced care as usual (Active Comparator): Participants receive a paper-based self-advocacy guide.
  Interventions: Behavioral: Enhanced Care as Usual

INTERVENTIONS:
Behavioral: Strong Together serious game — The Strong Together serious game program is an interactive, immersive education program in which participants quickly learn the behaviors of self-advocacy and the potential consequences of self-advocating or not. Participants receive weekly notifications for 12 weeks alerting them that a new serious game session is available and encourage them to complete one session per week.
  Arms: Serious game intervention
Behavioral: Enhanced Care as Usual — A self-advocacy patient brochure published by the National Coalition for Cancer Survivorship. This guide is not a part of usual care, but is freely available on the Internet.
  Arms: Enhanced care as usual

SUMMARY:
Individuals with cancer must overcome multiple, ongoing challenges ("self-advocate") related to their cancer experience to receive patient-centered care. Women with metastatic cancer often face significant challenges managing their quality of life concerns and cancer- and treatment-related symptoms. If they do not self-advocate to manage these concerns, they risk having poor quality of life, high symptom burden, and care that is not patient-centered. Serious games (video games that teach) are effective health interventions that allow users to vicariously engage in situations reflecting their personal experiences, receive meaningful information, and learn personally relevant skills that they can apply in real life.

The goal of the current study is to test the efficacy of a novel intervention using a serious game platform to teach self-advocacy skills to women with advanced cancer. The Strong Together intervention consists of a multi-session, interactive serious game application with tailored self-advocacy goal-setting and training. The serious game is based on a self-advocacy conceptual framework and applies behavior change theories and serious game mechanisms to promote skill development and implementation. The game works by immersing users in the experiences of characters who are women with advanced cancer; requiring users to make decisions about how the characters self-advocate; demonstrating the positive and negative consequences of self-advocating or not, respectively; and providing multiple, individualized feedback mechanisms and game features to enforce self-advocacy skill acquisition and transference to real life.

DETAILED DESCRIPTION:
Patient-centered care (e.g., incorporating patient preferences, needs, and values into all care aspects) is an essential component of high-quality care, associated with improved patient health, well-being, treatment adherence, and care coordination. Patients cannot participate in patient-centered care if they do not have the skills to self-advocate. Self-advocacy is defined as the ability to overcome health challenges by making informed healthcare decisions, communicating effectively with healthcare providers, and gaining strength through connection to others. Our work established that self-advocacy is associated with higher quality of life, lower symptom burden, higher patient-centered care, and fewer hospital admissions and emergency visits. Self-advocacy is particularly necessary in the advanced cancer setting where patients face numerous health challenges including complex treatment decisions, multiple cancer- and treatment-related symptoms, and poor quality of life. However, many patients struggle to self-advocate because they have not previously needed these skills or do not know how to apply these skills within their cancer experience. Interventions to teach patients self-advocacy are lacking, and the few programs that exist rely on non-interactive patient education that does not leverage behavior change or educational theories. There is a critical need for theoretically grounded interventions to teach patients with advanced cancer self-advocacy skills so that they can address health challenges related to their care and experience improved outcomes.

Technology-based serious games (educational video games) allow users to vicariously engage in situations reflecting their personal experiences, receive meaningful information, and learn personally relevant skills that they can apply in real life. Serious games are an ideal platform for teaching self-advocacy skills because they use immersive, motivational elements and mechanisms to provide highly-relevant skills-training. Serious games improve patient knowledge and skills though their mechanisms of action remain unclear.

Our team developed the Strong Together intervention which teaches self-advocacy skills in a serious game platform. Patients vicariously respond to health challenges managing symptoms, communicating with providers, and managing their health and are then exposed to the positive and negative consequences of self-advocating or not, respectively. It is based on our team's self-advocacy conceptual model, grounded in behavior change and educational theories, and integrates multiple mechanisms to promote learning outcomes. Our valid, reliable self-report self-advocacy measure captures the three dimensions of self-advocacy: informed decision-making, strength through connection, and effective communication. Our pilot randomized clinical trial (RCT) of the Strong Together intervention among N=70 women newly diagnosed with advanced breast or gynecologic cancer demonstrated feasibility (82% completed 6-month surveys, 71% engaged in all intervention sessions) and intervention acceptability (97% satisfied; 90% saw it as useful).

In the current study, the investigators will test the efficacy of the Strong Together intervention compared with an enhanced care as usual group in a larger, more diverse sample of women with advanced cancer.

ELIGIBILITY:
Inclusion Criteria:

* Female
* ≥18 years
* Diagnosed with advanced solid organ cancer within the past 6 months being treated with non-curative intent
* Have at least a 6-month life expectancy (as determined by their oncologist)
* Eastern Cooperative Oncology Group performance score of 0 to 2 (per health record or oncologist)
* Able to read and write in English

Exclusion Criteria:

* On hospice at the time of recruitment
* Impaired cognition (per health record)
* Other active, unstable mental health disorder

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Inclusion criteria are based on self-reported gender identity
Enrollment: 336 (Estimated)
Dates: Start 2022-08-22 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Mean change from baseline in self-advocacy scores on the Female Self-Advocacy in Cancer Survivorship (FSACS) Scale at 3 months | Baseline and 3 months
  The Female Self-Advocacy in Cancer Survivorship (FSACS) Scale is a 20-item, 6-point Likert-type scale (score range: 20-120). The scale is a validated measure of a woman with cancer's ability to engage in informed decision-making, strength through connection, and effective communication with healthcare providers. Higher scores indicate higher self-advocacy.
Mean change from baseline in self-advocacy scores on the Female Self-Advocacy in Cancer Survivorship (FSACS) Scale at 6 months | Baseline and 6 months
  The Female Self-Advocacy in Cancer Survivorship (FSACS) Scale is a 20-item, 6-point Likert-type scale (score range: 20-120). The scale is a validated measure of a woman with cancer's ability to engage in informed decision-making, strength through connection, and effective communication with healthcare providers. Higher scores indicate higher self-advocacy.

SECONDARY OUTCOMES:
Mean change from baseline in quality of life scores on the Functional Assessment of Cancer Therapy - General (FACT-G) Scale at 3 months | Baseline and 3 months
  The Functional Assessment of Cancer Therapy - General (FACT-G) is a 27-item, 5-point Likert-type scale (score range: 0-108). This scale captures physical, functional, social, and emotional well-being among patients with cancer. Higher scores indicate higher quality of life.
Mean change from baseline in quality of life scores on the Functional Assessment of Cancer Therapy - General (FACT-G) Scale at 6 months | Baseline and 6 months
  The Functional Assessment of Cancer Therapy - General (FACT-G) is a 27-item, 5-point Likert-type scale (score range: 0-108). This scale captures physical, functional, social, and emotional well-being among patients with cancer. Higher scores indicate higher quality of life.
Mean change from baseline in symptom burden scores on the M.D. Anderson Symptom Inventory (MDASI) at 3 months | Baseline and 3 months
  The M.D. Anderson Symptom Inventory (MDASI) is a 19-item, 11-point Likert-type scale consisting of two subscales (score range: 0-190. The first subscale assesses symptom severity of 13 common cancer- and treatment-related symptoms on a scale of 0 to 10. Higher scores indicate higher symptom severity. The second subscale assesses the degree to which symptoms interfere with daily life on a scale of 0 to 10. Higher scores indicate higher symptom interference.
Mean change from baseline in symptom burden scores on the M.D. Anderson Symptom Inventory (MDASI) at 6 months | Baseline and 6 months
  The M.D. Anderson Symptom Inventory (MDASI) is a 19-item, 11-point Likert-type scale consisting of two subscales (score range: 0-190. The first subscale assesses symptom severity of 13 common cancer- and treatment-related symptoms on a scale of 0 to 10. Higher scores indicate higher symptom severity. The second subscale assesses the degree to which symptoms interfere with daily life on a scale of 0 to 10. Higher scores indicate higher symptom interference.
Mean change from baseline in patient-perceived patient-centeredness of care scores on the Patient Centeredness of Care Scale (PCCS) at 3 months | Baseline and 3 months
  The Patient Centeredness of Care Scale (PCCS) is 14-item, 4-point Likert-type scale (score range: 0-42). This measure assesses patient perceptions of how patient-centered their oncologist interactions are, including the degree the oncologist explores the patient's health and illness experiences and finds common ground.
Mean change from baseline in patient-perceived patient-centeredness of care scores on the Patient Centeredness of Care Scale (PCCS) at 6 months | Baseline and 6 months
  The Patient Centeredness of Care Scale (PCCS) is 14-item, 4-point Likert-type scale (score range: 0-42). This measure assesses patient perceptions of how patient-centered their oncologist interactions are, including the degree the oncologist explores the patient's health and illness experiences and finds common ground.

OTHER OUTCOMES:
Changes from baseline in use of healthcare service utilization defined as hospital admissions, emergency room visits, and (un)planned clinic visits at 3 months | Baseline and 3 months
  Electronic Medical Record and self-report of the number of times the patient has gone to the Emergency Department, been admitted to a hospital, and had (un)scheduled clinic visits within the past three months
Changes from baseline in use of healthcare service utilization defined as hospital admissions, emergency room visits, and (un)planned clinic visits at 6 months | Baseline and 6 months
  Electronic Medical Record and self-report of the number of times the patient has gone to the Emergency Department, been admitted to a hospital, and had (un)scheduled clinic visits within the past three months
Intervention receipt | Baseline and 3 months
  Calculation of the time, duration, and intervention content used by participants.
Intervention mechanism usage | Baseline and 3 months
  Calculation of differences in primary and secondary outcome measures based on exposure to serious game mechanisms.
Intervention mechanism usage | Baseline and v6 months
  Calculation of differences in primary and secondary outcome measures based on exposure to serious game mechanisms.

CONTACTS AND LOCATIONS:
Locations (1):
- UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Thomas TH, Bender C, Rosenzweig M, Taylor S, Sereika SM, Babichenko D, You KL, Terry MA, Sabik LM, Schenker Y. Testing the effects of the Strong Together self-advocacy serious game among women with advanced cancer: Protocol for the STRONG randomized clinical trial. Contemp Clin Trials. 2023 Jan;124:107003. doi: 10.1016/j.cct.2022.107003. Epub 2022 Nov 13. PMID 36379436

DOCUMENTS (1):
  • Informed Consent Form (2023-12-06): https://cdn.clinicaltrials.gov/large-docs/76/NCT04813276/ICF_000.pdf